CLINICAL TRIAL: NCT04729959
Title: A Safety Run-In and Phase II Study Evaluating the Efficacy, Safety, and Impact on the Tumor Microenvironment of the Combination of Tocilizumab, Atezolizumab, and Fractionated Stereotactic Radiotherapy in Recurrent Glioblastoma
Brief Title: Testing the Addition of the Immune Therapy Drugs, Tocilizumab and Atezolizumab, to Radiation Therapy for Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-00410; NCI-2021-00410 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN010 (Other: NRG Oncology); NRG-BN010 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Astrocytoma, IDH-Wildtype; Recurrent Glioblastoma
MeSH Terms: conditions — Astrocytoma; Glioblastoma | interventions — atezolizumab; Specimen Handling; Magnetic Resonance Spectroscopy; tocilizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (tocilizumab, atezolizumab, FSRT) (Experimental): Patients receive systemic treatment with tocilizumab IV over 60 minutes with or without atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3 fractions over 3-5 days in the absence of disease progression or unacceptable toxicity. Starting 4 weeks from the first dose of systemic treatment, patients resume treatment with tocilizumab with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial.
  Interventions: Biological: Atezolizumab; Radiation: Fractionated Stereotactic Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Tocilizumab
- Group II, Arm I (tocilizumab, atezolizumab, FSRT, surgery) (Experimental): Patients receive systemic treatment with tocilizumab IV over 60 minutes with or without atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3 fractions over 3-5 days. Within 7-14 days after FSRT, patients undergo surgery. Within 21-24 days from the first dose of systemic treatment, patients resume treatment with tocilizumab with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial, as well as blood sample and tumor tissue collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Conventional Surgery; Radiation: Fractionated Stereotactic Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Tocilizumab
- Group II, Arm II (tocilizumab, atezolizumab, FSRT, surgery) (Experimental): Patients receive systemic treatment with atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3-5 fractions over 3-5 days. Within 7-14 days after FSRT, patients undergo surgery. Within 21-42 days from the first dose of systemic treatment, patients resume treatment with tocilizumab IV over 60 minutes with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo MRI and tumor tissue collection on study. Patients undergo MRI throughout the trial, as well as blood sample and tumor tissue collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Conventional Surgery; Radiation: Fractionated Stereotactic Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Tocilizumab

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Procedure: Biospecimen Collection — Undergo blood sample and tumor tissue collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Group II, Arm I (tocilizumab, atezolizumab, FSRT, surgery); Group II, Arm II (tocilizumab, atezolizumab, FSRT, surgery)
Procedure: Conventional Surgery — Undergo surgery
  Arms: Group II, Arm I (tocilizumab, atezolizumab, FSRT, surgery); Group II, Arm II (tocilizumab, atezolizumab, FSRT, surgery)
Radiation: Fractionated Stereotactic Radiation Therapy — Undergo FSRT
  Other Names: Fractionated Stereotactic Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Tocilizumab — Given IV
  Other Names: Actemra; IL-6 receptor monoclonal antibodies: tocilizumab; Immunoglobulin G1, Anti-(Human Interleukin 6 Receptor) (Human-Mouse Monoclonal MRA Heavy Chain), Disulfide with Human-Mouse Monoclonal MRA Kappa-Chain, Dimer; MRA; R-1569; RoActemra

SUMMARY:
This phase II trial studies the best dose and effect of tocilizumab in combination with atezolizumab and stereotactic radiation therapy in treating glioblastoma patients whose tumor has come back after initial treatment (recurrent). Tocilizumab is a monoclonal antibody that binds to receptors for a protein called interleukin-6 (IL-6), which is made by white blood cells and other cells in the body as well as certain types of cancer. This may help lower the body's immune response and reduce inflammation. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Fractionated stereotactic radiation therapy uses special equipment to precisely deliver multiple, smaller doses of radiation spread over several treatment sessions to the tumor. The goal of this study is to change a tumor that is unresponsive to cancer therapy into a more responsive one. Therapy with fractionated stereotactic radiotherapy in combination with tocilizumab may suppress the inhibitory effect of immune cells surrounding the tumor and consequently allow an immunotherapy treatment by atezolizumab to activate the immune response against the tumor. Combination therapy with tocilizumab, atezolizumab and fractionated stereotactic radiation therapy may shrink or stabilize the cancer better than radiation therapy alone in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum-tolerated dose (MTD) among three sequential dose levels: single-agent tocilizumab 4 mg/kg, single-agent tocilizumab 8 mg/kg, and tocilizumab 8 mg/kg + atezolizumab 1680 mg (each administered with fractionated stereotactic radiation therapy [FSRT]), to be used for subsequent phase II testing. (Safety Run-In) II. To determine the efficacy of the combination of tocilizumab (anti-IL6R), atezolizumab (anti-PD-L1), and FSRT in recurrent glioblastoma (GBM), as measured by the objective radiographic response rate (ORR). (Phase II [Non-Surgical Cohort])

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) in patients with recurrent GBM treated with the combination of tocilizumab (anti-IL6R) and FSRT (and atezolizumab [anti-PD-L1], if dose level 3 is MTD). (Phase II Non-Surgical Cohort and Safety Run-in Cohort) II. To estimate the overall survival (OS) in patients with recurrent GBM treated with the combination of tocilizumab (anti-IL6R) and FSRT (and atezolizumab [anti-PD-L1], if dose level 3 is MTD)), atezolizumab (anti-PD-L1), and FSRT. (Phase II Non-Surgical Cohort and Safety Run-in Cohort) III. To estimate the progression-free survival (PFS) in patients with recurrent GBM treated with the combination of tocilizumab (anti-IL6R), atezolizumab (anti-PD-L1), and FSRT. (Phase II Surgical Cohort) IV. To estimate the overall survival (OS) in patients with recurrent GBM treated with the combination of tocilizumab (anti-IL6R), atezolizumab (anti-PD-L1), and FSRT. (Phase II Surgical Cohort) V. To determine the rate and severity of adverse events (AEs) of the combination of tocilizumab (anti-IL6R), atezolizumab (anti-PD-L1), and FSRT in recurrent glioblastoma according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. (Separately in the Nonsurgical and Surgical Cohorts)

EXPLORATORY OBJECTIVES:

I. To determine the effect of the combination of atezolizumab (anti-PD-L1) and FSRT, with versus (vs.) without tocilizumab (anti-IL6R), on the GBM immune microenvironment. (Phase II Surgical Cohort) II. To evaluate the pharmacodynamic impact of the combination of tocilizumab (anti-IL6R), atezolizumab (anti-PD-L1), and FSRT on peripheral blood immune cell populations. (Phase II Surgical Cohort) III. To detect tumor and/or blood biomarkers associated with the outcomes of OS, PFS, and/or ORR in patients with recurrent GBM treated with the combination of tocilizumab (anti-IL6R), atezolizumab (anti-PD-L1), and FSRT. (Phase II Non-Surgical Cohort)

OUTLINE:

SAFETY RUN-IN: Patients receive systemic treatment with either tocilizumab intravenously (IV) over 60 minutes with or without atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3 fractions over 3-5 days. Starting 4 weeks from the first dose of systemic treatment, patients resume treatment with tocilizumab with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI) throughout the trial. (CLOSED TO ACCRUAL 08-AUG-2023)

GROUP I (NON-SURGICAL COHORT): Patients receive systemic treatment with tocilizumab IV over 60 minutes with or without atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3 fractions over 3-5 days in the absence of disease progression or unacceptable toxicity. Starting 4 weeks from the first dose of systemic treatment, patients resume treatment with tocilizumab with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial.

GROUP II (SURGICAL COHORT): Patients are randomized to 1 of 2 arms.

ARM I: Patients receive systemic treatment with tocilizumab IV over 60 minutes with or without atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3 fractions over 3-5 days. Within 7-14 days after FSRT, patients undergo surgery. Within 21-24 days from the first dose of systemic treatment, patients resume treatment with tocilizumab with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial, as well as blood sample and tumor tissue collection on study.

ARM II: Patients receive systemic treatment with atezolizumab IV over 30-60 minutes on day 1. Within 3-7 days, patients undergo FSRT for 3-5 fractions over 3-5 days. Within 7-14 days after FSRT, patients undergo surgery. Within 21-42 days from the first dose of systemic treatment, patients resume treatment with tocilizumab IV over 60 minutes with or without atezolizumab. Treatment repeats every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo MRI throughout the trial, as well as blood sample and tumor tissue collection on study.

After completion of study treatment, patients are followed up at 30 days, 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma, OR molecular diagnosis of glioblastoma per Consortium to Inform Molecular and Practical Approaches to Central Nervous System Tumor Taxonomy (c-IMPACT-NOW) criteria ("diffuse astrocytic glioma, IDH-wildtype, with molecular features of glioblastoma, World Health Organization [WHO] grade IV"; this requires presence of amplification of EGFR, whole chromosome 7 gain AND whole chromosome 10 loss, or TERT promoter mutation)
* Tumor that is in first recurrence following prior first-line radiation therapy (prior dose >= 40 Gy)

  * Note: Prior temozolomide, prior tumor-treating fields, and/or Gliadel wafers (if placed at initial tumor resection) are allowed, but none of these are required
* Unequivocal radiographic evidence of tumor progression by contrast-enhanced magnetic resonance imaging (MRI) scan within 21 days prior to registration
* Per radiation oncologist review of MRI within 21 days prior to registration, must have focus of progressive, contrast-enhancing tumor that is amenable to FSRT, defined as the following:

  * At least 1 cm x 1 cm contrast-enhancing tumor that is no greater than 4 cm in largest dimension
  * FSRT target is at least 0.5 cm from the optic chiasm and brainstem
  * Note, multifocal disease (i.e., other sites of tumor beyond the tumor being targeted for FSRT) is allowed if the above criteria are met for the tumor that is the proposed target for FSRT
* Surgical cohort only (Phase II only):

  * Must be a candidate for repeat surgery (significant debulking or gross total resection of the contrast enhancing area) as determined by the neurosurgeon or multidisciplinary team
* Tumor O-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) methylation status must be available from any prior GBM tumor specimen; results of routinely used methods for MGMT methylation testing (e.g. mutagenically separated polymerase chain reaction [MSPCR] or quantitative polymerase chain reaction [PCR]) are acceptable)
* The following intervals from previous treatments to registration are required to be eligible:

  * If prior radiation was < 60 Gy, an interval of at least 12 weeks (84 days) must have elapsed since the completion of radiation therapy
  * If prior radiation was >= 60 Gy, an interval of least 6 months (182 days) must have elapsed since the completion of radiation therapy, unless the target lesion for FSRT is outside of the 80% isodose line of the original radiation plan
  * At least 21 days from temozolomide
  * At least 28 days from any investigational (not Food and Drug Administration [FDA]-approved for glioblastoma) agents, or within a time interval less than at least 5 half-lives of the investigational agent whichever is shorter (Note: anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapeutic antibody or pathway-targeting agents are not allowed)
* Age >= 18 years
* Karnofsky performance status >= 70 within 14 days prior to registration
* History/physical examination within 14 days prior to registration
* Leukocytes >= 2,500/mm^3 (within 14 days prior to registration)
* Absolute neutrophil count >= 1,500/mm^3 (within 14 days prior to registration)
* Absolute lymphocyte count >= 800/mm^3 (within 14 days prior to registration)
* Platelets >= 100,000/mm^3 (within 14 days prior to registration)
* Hemoglobin >= 8 g/dL (within 14 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x ULN (within 14 days prior to registration)
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x ULN (within 14 days prior to registration)
* Alkaline phosphatase =< 2.5 x ULN (within 14 days prior to registration)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault (within 14 days prior to registration)
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of receipt of study treatment, and for 60 days (males) or 90 days (females) from the last dose of tocilizumab and for 5 months (150 days) after the last dose of atezolizumab. Administration of atezolizumab or tocilizumab may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to registration
* Patients positive for human immunodeficiency virus (HIV) are allowed on study (note: HIV testing is not required), but HIV-positive patients must have:

  * An undetectable viral load within 6 months of registration
  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

  * Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B
* For patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV ribonucleic acid [RNA]) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Availability of prior radiotherapy treatment plan details in Digital Imaging and Communications in Medicine (DICOM) format

Exclusion Criteria:

* Known somatic tumor mutation in IDH1 or IDH2 gene. If not previously completed, sequencing of the IDH1 and IDH2 genes is not required to determine trial eligibility
* Known germline DNA repair defect (mismatch repair deficiency, POLE mutation, e.g.). If not previously completed, germline sequencing is not required to determine trial eligibility
* Diffuse leptomeningeal disease
* Known contrast-enhancing tumor in brainstem or spinal cord. If not previously completed, spinal imaging is not required to determine trial eligibility
* Patients with clinically significant mass effect or midline shift (e.g., 1-2 cm of midline shift)
* Prior bevacizumab therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are excluded from this trial. Otherwise, patients with prior or concurrent malignancy are eligible
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon [IFN]-alpha or interleukin [IL]-2) within 4 weeks prior to registration
* Treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to registration
* Systemic corticosteroids used to treat brain edema and/or related symptoms at a dose of > 2 mg of dexamethasone (or equivalent) daily within 5 days prior to registration. Patients receiving systemic corticosteroids for other indications are excluded
* Patients with increased risk for gastrointestinal perforations including history of diverticulitis
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis.

  * Note: patients with the below conditions are eligible:

    * Autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible.
    * Controlled type 1 diabetes mellitus on a stable insulin regimen are eligible.
    * Eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only are permitted provided that they meet the following conditions:

      * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
      * Rash must cover less than 10% of body surface area (BSA)
      * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, fluocinolone 0.01%, desonide 0.05%, alclometasone dipropionate 0.05%)
      * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), or organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.)

  * Note: History of radiation pneumonitis in a prior radiation field (fibrosis) is permitted
* Patients with active tuberculosis (TB) are excluded
* Severe infections within 3 weeks prior to registration including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 1 week prior to registration
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to registration

  * Note: Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 21 days prior to registration or anticipation of need for a major surgical procedure during the course of study treatment
* Administration of a live, attenuated vaccine within 4 weeks before registration or anticipation that such a live, attenuated vaccine will be required during receipt of study treatment and up to 5 months after the last dose of study drug
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or nursing (and unwilling to discontinue) are excluded from this study. Atezolizumab and tocilizumab are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atezolizumab and tocilizumab breastfeeding should be discontinued if the mother is treated with atezolizumab and tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (Safety Run-In) | Up to 1 post-fractionated stereotactic radiation therapy (FRST) cycle of systemic therapy for which dose-limiting toxicity is reached (1 cycle = 4 weeks)
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0.
Maximum-tolerated dose (Safety Run-In) | Up to 1 post-FRST cycle of systemic therapy for which dose-limiting toxicity is reached (1 cycle = 4 weeks)
Objective radiographic response rate (Phase II, Non-Surgical Cohort) | Up to 6 months from enrollment
  Will be determined using modified Response Assessment in Neuro-oncology with the pretreatment magnetic resonance imaging as baseline. Frequencies and percent of responses will be provided for patients with measurable disease.

SECONDARY OUTCOMES:
Progression-free survival (PFS) (Phase II, Non-Surgical Cohort) | Time from study enrollment to disease progression or death from any cause, assessed up to 2 years
  PFS curves will be assessed via the Kaplan-Meier method.
Overall survival (Phase II, Non-Surgical Cohort) | From study enrollment to death from any cause, assessed up to 2 years
  Will be assessed via the Kaplan-Meier method.
Progression-free survival (Phase II, Non-Surgical Cohort) | From randomization to disease progression or death from any cause, assessed up to 2 years
  Kaplan-Meier method will be used to estimate the PFS within each randomized arm separately as well as combined.
Overall survival (Phase II, Surgical Cohort) | From study enrollment to death from any cause, assessed up to 2 years
  Will be assessed via the Kaplan-Meier method.
Incidence of adverse events (Surgical Cohort and Non-Surgical Cohort) | Up to 2 years
  Will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Comprehensive summaries of all adverse events by treatment arm will be generated and examined. Counts and frequencies of worst (highest score) adverse event per patient will be presented overall and by adverse event type category, separately by assigned treatment group. The proportion of patients with at least one grade 3 or higher adverse event will be compared between treatment arm. Similarly, frequencies for specific potentially treatment related adverse events where grade 3 or higher events are noted may be compared. Any frequencies to be tested will be evaluated using the chi-square or exact test as appropriate, with two-sided significance level 0.05.

OTHER OUTCOMES:
Immune response (Phase II, Surgical Cohort) | Baseline and cycle 2, day 1 (1 cycle = 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bagley, Principal Investigator — NRG Oncology
Locations (110):
- United States (110):
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Renown Regional Medical Center, Reno, Nevada
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT04729959/SAP_000.pdf
  • Informed Consent Form (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT04729959/ICF_001.pdf